CLINICAL TRIAL: NCT01758042
Title: Combined Haploidentical Reduced Intensity Bone Marrow and Kidney Transplantation for Patients With Chronic Kidney Disease and Advanced Hematological Disorders
Brief Title: Bone Marrow and Kidney Transplant for Patients With Chronic Kidney Disease and Blood Disorders
Acronym: BMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Director of Clinical Research, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001355
Record Dates: First submitted 2012-12-17; First posted 2012-12-31 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Disease; Acute Myeloid Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Chronic Myelogenous Leukemia (CML); Chronic Lymphocytic Leukemia (CLL); Non-Hodgkin's Lymphoma (NHL); Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndrome (MDS); Aplastic Anemia; AL Amyloidosis; Diamond Blackfan Anemia; Myelofibrosis; Myeloproliferative Disease; Sickle Cell Anemia; Autoimmune Diseases; Thalassemia
Keywords: Kidney; Chronic Kidney Disease; CKD; Bone Marrow; Bone Marrow Transplant; BMT; Leukemia; AML; ALL; CML; CLL; MM; NHL; MDS
MeSH Terms: conditions — Renal Insufficiency, Chronic; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndromes; Anemia, Aplastic; Immunoglobulin Light-chain Amyloidosis; Anemia, Diamond-Blackfan; Primary Myelofibrosis; Myeloproliferative Disorders; Anemia, Sickle Cell; Autoimmune Diseases; Thalassemia; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical Bone Marrow/Kidney (Other): Single Arm Study
  Interventions: Procedure: Haploidentical Bone Marrow/Kidney

INTERVENTIONS:
Procedure: Haploidentical Bone Marrow/Kidney — Combined bone marrow and kidney transplantation using a haploidentical donor.

SUMMARY:
The main purpose of this study is to examine the outcome of a combined bone marrow and kidney transplant from a partially matched related (haploidentical or "haplo") donor. This is a pilot study, you are being asked to participate because you have a blood disorder and kidney disease. The aim of the combined transplant is to treat both your underlying blood disorder and kidney disease. We expect to have about 10 people participate in this study.

Additionally, because the same person who is donating the kidney will also be donating the bone marrow, there may be a smaller chance of kidney rejection and less need for long-term use of anti-rejection drugs.

Traditionally, very strong cancer treatment drugs (chemotherapy) and radiation are used to prepare a subject's body for bone marrow transplant. This is associated with a high risk for serious complications, even in subjects without kidney disease. This therapy can be toxic to the liver, lungs, mucous membranes, and intestines. Additionally, it is believed that standard therapy may be associated with a higher risk of a complication called graft versus host disease (GVHD) where the new donor cells attack the recipient's normal body. Recently, less intense chemotherapy and radiation regimens have been employed (these are called reduced intensity regimens) which cause less injury and GVHD to patients, and thus, have allowed older and less healthy patients to undergo bone marrow transplant. In this study, a reduced intensity regimen of chemotherapy and radiation will be used with the intent of producing fewer toxicities than standard therapy.

Typical therapy following a standard kidney transplant includes multiple lifelong medications that aim to prevent the recipient's body from attacking or rejecting the donated kidney. These are called immunosuppressant drugs and they work by "quieting" the recipient's immune system to allow the donated kidney to function properly. One goal in our study is to decrease the duration you will need to be on immunosuppressant drugs following your kidney transplant as the bone marrow transplant will provide you with the donor's immune system which should not attack the donor kidney.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-70
* Underlying hematological disorder which is potentially curable with allogeneic bone marrow transplantation. This includes, but is not limited to: acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myelogenous leukemia (CML), chronic lymphocytic leukemia (CLL), non-Hodgkin lymphoma (NHL), Hodgkin lymphoma, multiple myeloma (MM), myelodysplastic syndrome (MDS), AL amyloidosis, diamond blackfan anemia, myelofibrosis or other myeloproliferative disease, sickle cell anemia, and thalassemia.
* Existence of haploidentical first degree relative who passes standard donor evaluations for bone marrow and kidney donation
* LVEF > 40% as measured by echocardiography or MUGA
* FEV1, FVC, and DLCO > 50% of predicted as measured by standard PFTs
* Total bilirubin < 2.0 (unless diagnosis of Gilbert's or hemolysis is made) and AST, ALT, alkaline phosphatase all < 5x institutions upper limit of normal
* ABO compatibility in the host vs. graft direction
* Men and women of reproductive potential must agree to use a reliable method of birth control during the treatment, and women should do so for a period of 1 year following the transplant.
* Participants should be on dialysis or have an estimated or measured CrCl < 35 ml/min
* Life expectancy greater than six months.
* Recipient ability to understand and provide informed consent

Exclusion Criteria:

* Active serious infection
* Participation in other investigational drug use at the time of enrollment
* Contraindication to therapy with any one of the proposed agents (e.g., history of allergy to rabbit serum in ATG)
* Serologic positivity for HIV, HCV, or HbsAg positivity
* ABO blood group incompatibility in the host-vs-graft direction
* Active serious infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-11; Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who die of treatment-related complications. | 100 days and 1 year post transplant
  Assess safety of haploidentical combined bone marrow and kidney transplantation as measured treatment related mortality.

SECONDARY OUTCOMES:
Number of patients with acute and delayed renal allograft rejection | 2 years post-transplant

OTHER OUTCOMES:
Number of patients who are able to discontinue immunosuppressive therapy by one year post transplant | one year post transplant
Number of patients who develop acute and chronic graft versus host disease (GVHD). | post transplant
Number of patients who relapse from their underlying hematological disease | 6 months, 1 year, and 2 years post transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin A Chen, M.D., Principal Investigator — Director of Clinical Research, Massachusetts General Hospital Bone Marrow Transplant Program
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chen YB, Elias N, Heher E, McCune JS, Collier K, Li S, Del Rio C, El-Jawahri A, Williams W, Tolkoff-Rubin N, Fishman JA, McAfee S, Dey BR, DeFilipp Z, O'Donnell PV, Cosimi AB, Sachs D, Kawai T, Spitzer TR. Haploidentical hematopoietic cell and kidney transplantation for hematological malignancies and end-stage renal failure. Blood. 2019 Jul 11;134(2):211-215. doi: 10.1182/blood.2019000775. Epub 2019 May 31. PMID 31151984